CLINICAL TRIAL: NCT00575640
Title: Hydralazine as a Demethylating Agent in Rectal Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No enrollment
Sponsor: University of Arkansas (Other)
Responsible Party: Ahmed M. Safar, MD, University of Arkansas for Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2004-03
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Hydralazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): The objective of this study is to determine the MTD for Hydralazine added to standard neoadjuvant chemotherapy for operable recta cancer. Four dose levels of hydralazine are planned:
  Dose Level 1: 150 mg/d 50 mg PO TID Dose Level 2: 200 mg/d 50 mg PO QID Dose Level 3: 225 mg/d 75 mg PO TID
  Interventions: Drug: Hydralazine

INTERVENTIONS:
Drug: Hydralazine — Dose Level 1: 150 mg/d 50 mg PO TID Dose Level 2: 200 mg/d 50 mg PO QID Dose Level 3: 225 mg/d 75 mg PO TID

SUMMARY:
Clinically feasible dose of Hydralazine for ~ 3 months, by virtue of its demethylating effect, will:

1. Result in re-expression of epigenetically silenced TSGs in rectal cancer specimens.
2. Decrease the global methylation in primary cancer cells compared to pre-treatment

DETAILED DESCRIPTION:
This study will be conducted as a phase I/II clinical trial. In addition to determining the maximum tolerated dose (MTD) of hydralazine, the phase I trial will be performed to identify unexpected toxicities that may occur when hydralazine is used in conjunction with neoadjuvant chemotherapy in normotensive patients with rectal cancer. Once the phase I trial is successfully completed, the phase II trial to evaluate the efficacy of hydralazine in producing a demethylation effect will begin.

This phase I/II trial will require between 31 to 47 patients to complete.

• Phase I Study

The objective of this study is to determine the MTD for Hydralazine added to standard neoadjuvant chemotherapy for operable recta cancer. Four dose levels of hydralazine are planned:

Dose Level 1: 150 mg/d 50 mg PO TID Dose Level 2: 200 mg/d 50 mg PO QID Dose Level 3: 225 mg/d 75 mg PO TID

ELIGIBILITY:
Inclusion Criteria:

The principal objective of this study is to perform a molecular evaluation for the reversal of methylation in clinical material collected at two different time points. The first sample representing untreated (the biopsy sample), and later a hydralazine-treated specimen (the resection specimen). Accordingly, we are not using routine inclusion criterion for enrollment (such as histology or clinical stage), but realize that the majority of operable rectal cancers will be stages II-III, and that treatment-again not specified or restricted-will very likely follow the standard therapy for this disease (infusional 5-Fluorouracil and radiation therapy). The accrual target at the phase II segment of this trial is small and that does not allow for any traditional clinical endpoints assessment (such as response rate, time to treatment failure or survival). Accordingly, we do not plan on following these endpoint as part of this study.

Patients referred to the surgery or gastroenterology services for diagnostic evaluation for rectal cancer will be candidates to participate in this study. Patients with history of elevated blood pressure and who are already on anti-hypertensive drugs would be ideal candidates for this project. In such situation, hydralazine will replace other anti-hypertensives for the duration of study only. There is no age limit for this study. Inclusion criteria are as follows:

1. Operable rectal cancer (the overwhelming majority are Adenocarcinoma)
2. Signed informed consent
3. Baseline blood pressure OFF anti-hypertensives over 100/50 mmHg

Exclusion Criteria:

1. Pre-existing hypotension (as defined in this protocol BP 100/50)
2. Pre-existing liver disease (liver function tests over 2x upper limits of normal ULM).
3. Pre-existing kidney (serum creatinine over 2 mg/dl).
4. Medical necessity to remain on beta-blockers that cannot be met by other agents.
5. Coronary even in the preceding 2 months prior to enrollment. Coronary evens include any of the following:

   * Acute Myocardial Infarction
   * Cardiac catheterization regardless of outcome of procedure or need of intervention
   * History of Valvular heart disease
   * History of hypertrophic cardiomyopathy with left ventricular outflow tract obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-11; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The study design calls for an initial phase of dose-escalation in cohorts of 3 patients. There are no intra-patient changes in dose.

SECONDARY OUTCOMES:
Subsequent to this Phase I scheme, the study will continue with the selected dose-level (on toxicity and tolerability grounds) to accrue patients in a phase II scheme.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Safar, MD, Principal Investigator — University of Arkansas